CLINICAL TRIAL: NCT01973829
Title: The Checklist for Early Recognition and Treatment of Acute Illness (CERTAIN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, CONS-CRITICAL CARE, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-007998
Record Dates: First submitted 2013-10-23; First posted 2013-11-01 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Critical Illness; Sepsis; Respiratory Failure; Shock; Coma; Bleeding; Trauma
Keywords: CERTAIN, Checklist, ICU, Outcome, Adults
MeSH Terms: conditions — Critical Illness; Sepsis; Respiratory Insufficiency; Shock; Coma; Hemorrhage; Wounds and Injuries | interventions — Checklist; Association

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baseline arm (Other): baseline data (50 patients or 3 months per center)
  Interventions: Other: Checklist for Early Recognition and Treatment of Acute Illness (CERTAIN)

INTERVENTIONS:
Other: Checklist for Early Recognition and Treatment of Acute Illness (CERTAIN) — This study is about training and implementation of best critical care practices in the international ICUs with variable resources facilitated by access to a specifically designed electronic checklist
  Other Names: Checklist

SUMMARY:
The purpose of the study is to test whether the health care provider access and training in CERTAIN (Checklist for Early Recognition and Treatment of Acute Illness), would facilitate timely and error free best-practice delivery and minimize preventable death and costly complications in critically ill patients.

ELIGIBILITY:
Inclusion:

All adult (≥ 18 years) patients admitted for the first time to the participating ICUs will be included.

Exclusion:

Not critically Ill, admitted for low risk monitoring, planned ICU admissions for routine postoperative surveillance for less than 24 hours after uncomplicated surgery, readmission and transferred from outside ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5215 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Adherence to best critical care practices | Participants will be followed for the duration of ICU stay, an expected average of 2 weeks
  Adherence to best practice in initial evaluation and treatment of critically ill medical and surgical patients Appropriate shock resuscitation Appropriate sepsis treatment Appropriate mechanical ventilation Appropriate peptic ulcer, deep vein thrombosis and infectious disease prophylaxis
ICU and hospital lengths of stay | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Patient will be followed till they get discharged from hospital for whatever length they stay.

SECONDARY OUTCOMES:
Mortality for 4 weeks | Participants will be followed for the duration of 4 weeks and hospital discharge (up to 10 weeks post discharge)
  Patient will be followed for 4 weeks and hospital discharge(up to total 10 weeks post discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Ognjen Gajic, MD, Principal Investigator — Mayo Clinic; Marija Kojicic, MD, Principal Investigator — Institute for Pulmonary Diseases, Novi Sad, Serbia; Rahul Kashyap, MD, Study Director — Mayo Clinic; Marcus Schultz, MD, Principal Investigator — University of Amsterdam; Michelle N Gong, MD, Principal Investigator — Montefiore Medical Center, New York USA; Oguz Kilickaya, MD, Principal Investigator — Gulhane Military Medical Faculty, Ankara, Turkey; Neill Adhikari, MD, Principal Investigator — University of Toronto, Toronto Canada; Linda Bucher, PhD, Principal Investigator — College of Health Sciences, University of Delavere, Delawere USA; Daniel Talmor, MD, Principal Investigator — Beth Israel Deakoness Medical Center, Boston USA; Yue Dong, MD, Study Director — Mayo Clinic
Locations (30):
- Gomel Regional Clinical Hospital, Homyel, Belarus
- Bosnia and Herzegovina (3):
  - University Hospital Banja Luka, Banja Luka
  - Sveučilišna klinička bolnica, Mostar
  - Prim.Dr. Abdulah Nakaš, Sarajevo
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- China (7):
  - Beijing Hospital, Beijing
  - Guang An Men Hospital, Beijing
  - China West China Hospital, Chengdu
  - 1st Affiliated Hospital of Guangzhou Medical University, Guangzhusi
  - Anhui Province Hospital, Hefei
  - China Shanghai Changhai Hospital, Shanghai
  - Tianjin First Center Hospital, Tianjin
- KBC Rijeka, Rijeka, Croatia
- Centro De Diagnostica Imagenes Medicina Avanzada y Telemedicina CEDIMAT, Santo Domingo, Dominican Republic
- India (3):
  - Kasturba Hospital, Manial, Karnataka
  - Lok Nayak Hospital, New Delhi, National Capital Territory of Delhi
  - Ispat General Hospital, Raurkela, Odisha
- St James Hosptial, Dublin, Ireland
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ), Mexico City, Mexico
- Central State University Hospital, Ulaanbaatar, Mongolia
- Shaukat Khanum Memorial Cancer Hospital and Research Center, Lahore, Pakistan
- Philippines (2):
  - St. Luke's Medical Center, Manila
  - The Med City Hospital, Manila
- Heliodor Swiecicki Clinical Hospital at the Karol Marcinkowski Medical University in Poznań, Poznan, Poland
- King Abdulaziz Medical City,, Riyadh, Saudi Arabia
- Serbia (2):
  - Military Medical Academy, Belgrade
  - The Institute for pulmonary diseases of Vojvodina, Kamenitz
- Turkey (Türkiye) (2):
  - Akdeniz University Hospital, Antalya
  - Gulhane Military Medical Faculty, Antalya
- International hospital Kampala, Kampala, Uganda

REFERENCES:
- [Derived] Tekin A, Swart P, Flurin L, Vukoja M, Kashyap R, Schultz MJ, Gajic O, Dong Y; CERTAIN investigators of the Society of Critical Care Medicine Discovery Network. The Weekend Effect on Evidence-Based Care Adherence Before and After Implementation of Checklist-Based Care in the Intensive Care Unit: A Multinational Study. J Intensive Care Med. 2025 Nov 24:8850666251396016. doi: 10.1177/08850666251396016. Online ahead of print. PMID 41284657
- [Derived] Vukoja M, Dong Y, Adhikari NKJ, Schultz MJ, Arabi YM, Martin-Loeches I, Hache M, Gavrilovic S, Kashyap R, Gajic O; Checklist for Early Recognition and Treatment of Acute Illness and Injury (CERTAIN) Investigators of the SCCM Discovery Network. Checklist for Early Recognition and Treatment of Acute Illness and Injury: An Exploratory Multicenter International Quality-Improvement Study in the ICUs With Variable Resources. Crit Care Med. 2021 Jun 1;49(6):e598-e612. doi: 10.1097/CCM.0000000000004937. PMID 33729718
- See also: education and introduction website — http://icertain.org/